CLINICAL TRIAL: NCT07242599
Title: A Multicenter, Randomized, Open-label, Parallel-controlled, Event-driven, Blinded-endpoint Trial Evaluating the Efficacy and Safety of Ongericimab Injection in High-risk Stroke Patients With Intracranial or Extracranial Atherosclerotic Stenosis.
Brief Title: Ongericimab Injection Reducing Recurrence of Ischemic Stroke
Acronym: ORIS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Capital Medical University, Professor in Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORIS-2025-10
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Ischemic Cerebral Infarction
Keywords: ischemic stroke; lipid lowering therapy; Ongericimab Injection; LDL-C target
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (High target group) (Active Comparator): Standardized lipid-lowering therapy according to the Chinese Stroke Association Guidelines for Clinical Management of Cerebrovascular Diseases to achieve an LDL-C target below 70 mg/dL (1.8 mmol/L).
  Interventions: Combination Product: High target group
- Intervention group (Low target group) (Experimental): Ongericimab subcutaneous injection once every two weeks (150mg) or every four weeks(300mg) combined with standardized lipid-lowering therapy to achieve an LDL-C target below 55 mg/dL (1.4 mmol/L)
  Interventions: Combination Product: Low target group

INTERVENTIONS:
Combination Product: High target group — Standardized lipid-lowering therapy according to the Chinese Stroke Association Guidelines for Clinical Management of Cerebrovascular Diseases to achieve an LDL-C target below 70 mg/dL (1.8 mmol/L)
  Arms: Control group (High target group)
Combination Product: Low target group — Ongericimab subcutaneous injection once every two weeks (150mg) or every four weeks(300mg) combined with standardized lipid-lowering therapy to achieve an LDL-C target below 55 mg/dL (1.4 mmol/L)
  Arms: Intervention group (Low target group)

SUMMARY:
The Oris trial aims to evaluate whether the use of Ongericimab injection in patients with atherosclerotic ischemic cerebrovascular disease within 3 months of onset can reduce the risk of recurrent major cardiovascular events by achieving lower lipid-lowering target values (LDL-C < 1.4 mmol/L).

ELIGIBILITY:
Inclusion Criteria:

* Obtaining informed consent；
* Age ≥18 years；
* Patients with ischemic stroke within 3 months( NIHSS<15 before randomization);
* Presence of ≥50% stenosis in major intracranial or extracranial arteries, and related to the symptoms of the current episode or the location of infarction；
* LDL-C ≥ 70 mg/dL (1.8 mmol/L) at screening.

Exclusion Criteria:

* History of cerebral hemorrhage at any time (microhemorrhages present only on SWI are not an exclusion criterion)
* Hemorrhage or other pathological neurological conditions on baseline brain CT/MRI (e.g., vascular malformations, tumors, abscesses, or common non-ischemic brain diseases like multiple sclerosis);
* Presence of isolated sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness or vertigo, but no evidence of recent infarction on baseline head CT or MRI;
* Unable to complete the assessment of intracranial and extracranial arterial stenosis before randomization
* mRS score≥2 before onset (based on assessment of medical history);
* Stroke caused by angioplasty/vascular surgery;
* Cardioembolic stroke caused by atrial fibrillation, artificial heart valves, endocarditis, mitral stenosis, sinus node dysfunction, etc.
* Most recent fasting triglycerides >400 mg/dL (4.5 mmol/L) prior to randomization;
* Uncontrolled hypertension (SBP >180 mmHg or DBP >110 mmHg);
* Hypothyroidism diagnosed within 1 month before randomization.
* Severe renal impairment (eGFR <30 mL/min/1.73m²);
* Active liver disease or dysfunction (AST/ALT >3×ULN within 30 days pre-randomization);
* NYHA Class III/IV heart failure within 1 year prior to randomization;
* Life-limiting non-cardiovascular diseases (life expectancy <1 years);
* Malignancy within 10 years (excluding adequately treated basal cell carcinoma, cervical CIS, DCIS, or stage 1 prostate cancer);
* Active phase of infection (including respiratory tract infection, urinary tract infection, or gastroenteritis), or currently using or planning to use oral or intravenous anti-infective treatment due to infection;
* Known hypersensitivity to monoclonal antibody therapies;
* PCSK9 inhibitor use within 3 months before randomization.
* Participation in other drug/device trials within 30 days;
* History of severe drug or alcohol abuse within the past year.
* Women of childbearing potential without contraception, pregnancy, or lactation;
* Inability to understand or comply with the study due to mental illness, cognitive, or emotional disorders, or other reasons deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4398 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
The major cardiovascular events | A median of 2 years follow-up
  The composite primary end point of major cardiovascular events includes ischemic stroke, myocardial infarction, death from cardiovascular causes.

SECONDARY OUTCOMES:
New ischemic stroke | A median follow-up of 2 years
  Ischemic stroke refers to acute focal cerebral or retinal infarction, excluding other non-ischemic causes, and meeting any of the following conditions: (1) clinical symptoms or imaging evidence of acute new focal neurological deficit lasting more than 24 hours; or (2) focal symptoms or signs lasting less than 24 hours, but with imaging evidence of new infarction; or (3) progression of pre-existing vascular ischemic stroke (i.e., NIHSS increase of ≥ 4 on the basis of the primary ischemic stroke, excluding hemorrhagic transformation after infarction or symptomatic intracranial hemorrhage) lasting more than 24 hours, with new ischemic changes on head MRI or CT.
Myocardial infarction | A median of 2 year follow-up
Vascular death | A median of 2 years follow-up
Poor functional prognosis (mRS score > 1) at 1 year | A median of 2 years follow-up
Severity of new stroke | A median of 2 years follow-up
Absolute and percent changes in LDL-C levels | A median of 2 years follow-up
Absolute and percent changes in Lp(a) levels. | A median of 2 years follow-up
Treatment-emergent serious adverse events (SAEs) and adverse events (AEs) | A median of 2 years follow-up
  Treatment-emergent serious adverse events (SAEs) and adverse events (AEs) include cerebral hemorrhage, injection site infections, muscle-related adverse events, new-onset diabetes mellitus, and clinically significant laboratory abnormalities encompassing hepatic/renal function markers, creatine kinase (CK), fasting glucose, and glycated hemoglobin (HbA1c) during the double-blind treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Background] Turan TN, Nizam A, Lynn MJ, Egan BM, Le NA, Lopes-Virella MF, Hermayer KL, Harrell J, Derdeyn CP, Fiorella D, Janis LS, Lane B, Montgomery J, Chimowitz MI. Relationship between risk factor control and vascular events in the SAMMPRIS trial. Neurology. 2017 Jan 24;88(4):379-385. doi: 10.1212/WNL.0000000000003534. Epub 2016 Dec 21. PMID 28003500
- [Result] Shao C, Zhang S, Cheng Z, Yang K, Wang G, Shi X, Yang H, Ji Y, Li H, Zhang S, Ma J, Pei Z, Zhang Y, Li Y, Li L, Zheng Y, Shao C, Zhang M, Hao Y, Tang YD. Efficacy and safety of ongericimab in Chinese statin-intolerant patients with primary hypercholesterolemia or mixed dyslipidemia: a randomized, placebo-controlled phase 3 trial. Atherosclerosis. 2025 Aug;407:120408. doi: 10.1016/j.atherosclerosis.2025.120408. Epub 2025 Jun 16. PMID 40543299
- [Result] Lin J, Ji Y, Wang G, Ma X, Yao Z, Han X, Chen J, Chen J, Huang W, Xu G, Peng D, Yan P, Qiao P, He Y, Tang Y, Wang M, Zhang M, Yu J, Hao Y, Ma C. Efficacy and safety of ongericimab in Chinese patients with heterozygous familial hypercholesterolemia: A randomized, double-blind, placebo-controlled phase 3 trial. Atherosclerosis. 2025 Apr;403:119120. doi: 10.1016/j.atherosclerosis.2025.119120. Epub 2025 Jan 29. PMID 39999660
- [Result] Xu YY, Chen WQ, Wang MX, Pan YS, Li ZX, Liu LP, Zhao XQ, Wang YL, Li H, Wang YJ, Meng X; CNSR-III Investigators. Lipid management in ischaemic stroke or transient ischaemic attack in China: result from China National Stroke Registry III. BMJ Open. 2023 Mar 8;13(3):e069465. doi: 10.1136/bmjopen-2022-069465. PMID 36889830
- [Result] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Result] Amarenco P, Bogousslavsky J, Callahan A 3rd, Goldstein LB, Hennerici M, Rudolph AE, Sillesen H, Simunovic L, Szarek M, Welch KM, Zivin JA; Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med. 2006 Aug 10;355(6):549-59. doi: 10.1056/NEJMoa061894. PMID 16899775
- [Result] Amarenco P, Kim JS, Labreuche J, Charles H, Abtan J, Bejot Y, Cabrejo L, Cha JK, Ducrocq G, Giroud M, Guidoux C, Hobeanu C, Kim YJ, Lapergue B, Lavallee PC, Lee BC, Lee KB, Leys D, Mahagne MH, Meseguer E, Nighoghossian N, Pico F, Samson Y, Sibon I, Steg PG, Sung SM, Touboul PJ, Touze E, Varenne O, Vicaut E, Yelles N, Bruckert E; Treat Stroke to Target Investigators. A Comparison of Two LDL Cholesterol Targets after Ischemic Stroke. N Engl J Med. 2020 Jan 2;382(1):9. doi: 10.1056/NEJMoa1910355. Epub 2019 Nov 18. PMID 31738483